CLINICAL TRIAL: NCT04120610
Title: FlowMet-R Blood Flow Measurement for the Diagnosis of Peripheral Artery Disease (PAD) and Critical Limb Ischemia (CLI)
Brief Title: FlowMet-R Blood Flow Measurement for the Diagnosis of Peripheral Artery Disease and Critical Limb Ischemia
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision to terminate study prior to reaching full sample size.
Sponsor: Medtronic Endovascular (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: 30081919
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Claudication; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy: Healthy cohort is an age-matched population (over 40 years old) without history of PAD or suspected PAD. Healthy cohort will receive FlowMet-R measurement, Ankle Brachial Index (ABI), and Toe Brachial Index (TBI) measurements.
  Interventions: Diagnostic Test: FlowMet-R; Diagnostic Test: ABI; Diagnostic Test: TBI
- Peripheral Artery Disease: PAD cohort is all-comers to the vascular lab that are scheduled to undergo assessment for Peripheral Artery Disease (PAD) or have a planned endovascular or surgical intervention to address PAD and will receive FlowMet-R measurement in addition to their routine standard of care.
  Interventions: Diagnostic Test: FlowMet-R; Diagnostic Test: ABI; Diagnostic Test: TBI

INTERVENTIONS:
Diagnostic Test: FlowMet-R — FlowMet-R is a noninvasive blood flow measurement.
Diagnostic Test: ABI — Ankle Brachial Index is a ratio-metric blood pressure measurement in the ankle and arm.
Diagnostic Test: TBI — Ankle Brachial Index is a ratio-metric blood pressure measurement in the toe and arm.

SUMMARY:
Non-randomized, multi-center, longitudinal study of healthy subjects and subjects with PAD who are scheduled for ABI, TBI, and either Duplex Ultrasound or Angiographic assessments in a vascular clinic.

DETAILED DESCRIPTION:
Patients scheduled for peripheral vascular examination and healthy controls will be measured with the FlowMet-R, a noninvasive blood flow monitor, and compared to gold standard diagnostics - ABI, TBI, and Doppler Ultrasound. Sensitivity and specificity of the FlowMet-R device output in diagnosing PAD and CLI will be assessed on initial visit, 3-month followup, and 6-month followup.

ELIGIBILITY:
Inclusion Criteria:

PAD Positive Cohort

* Subject meets PAD positive criteria
* Subject is willing and able to provide informed consent
* Subject is willing and able to comply with study procedures
* Subject is able to understand the study procedures
* Subject is scheduled for vascular examination that includes noninvasive assessments as standard of care: ABI, TBI, and either a Duplex Ultrasound or Angiogram

Healthy Cohort

* Subject is willing and able to provide informed consent.
* Subject is willing and able to comply with the study procedures.
* Subject is able to understand the study procedures.
* Subject has no history of positive PAD diagnosis, and is not currently suspected of having PAD.

Exclusion Criteria:

PAD Positive Cohort

* Subject is under 40 or unable to consent.
* Subject has any medical condition, which, in the judgment of the Investigator and/or designee, makes the subject a poor candidate for the investigational study.
* Subject is excluded from analysis if no stenosis is found during Doppler but Tibial disease is suspected and Tibial ultrasound is not able to be performed.
* Subject does not have a suitable finger to attach the FlowMet-R probe.
* Subject does not have a suitable 1st or 2nd digit to attach FlowMet-R probe on the limb of interest.
* Subject has undergone revascularization within the last 90 days
* Subject cannot lay safely in a supine position.

Healthy Cohort

* Subject is under 40 or unable to consent.
* Subject has any medical condition, which, in the judgment of the Investigator and/or designee, makes the subject a poor candidate for the investigational study.
* One or more limbs has a prior or current diagnosis of PAD, or is reasonably suspected of having a diagnosis of PAD.
* Subject does not have a suitable finger to attach the FlowMet-R probe.
* Subject does not have a suitable 1st or 2nd digit to attach FlowMet-R probe.
* Subject has undergone revascularization within the last 90 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The PAD cohort population is persons who have known or suspected peripheral artery disease, and are being seen at a vascular clinic for evaluation.
  The Healthy cohort population is adult persons over 40 without history of PAD and who are not currently suspected of suffering from PAD.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Iowa Clinic, Des Moines, Iowa
  - Mercy Research, Chesterfield, Missouri
  - The Mt. Sinai Hospital, New York, New York
  - Ohio Health, Columbus, Ohio
  - Ascension Seton, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 205 subjects were consented in the study. Of the 205 subjects, 10 subjects were screen fails due to I/E criteria, resulting in 195 total subjects enrolled.
  There were limitations discovered in the study design during enrollment due to classification of PAD and CLI from respective sites. Patients were categorized based on observed ABI, TBI and Rutherford Classification regardless of enrollment cohort.
Units Other Than Participants: limbs
Groups:
- Healthy: Healthy cohort includes patients over 40 years old without history of PAD or suspected PAD, where the ABI>0.9 and ABI≤1.4 or TBI>0.7. Healthy cohort will receive FlowMet-R measurement, Ankle Brachial Index (ABI), and Toe Brachial Index (TBI) measurements.
  FlowMet-R: FlowMet-R is a noninvasive blood flow measurement.
  ABI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the ankle and arm.
  TBI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the toe and arm.
- Peripheral Artery Disease: PAD cohort is all-comers to the vascular lab that are scheduled to undergo assessment for Peripheral Artery Disease (PAD) or have a planned endovascular or surgical intervention to address PAD. PAD cohort patients will receive FlowMet-R measurement in addition to their routine standard of care.
  FlowMet-R: FlowMet-R is a noninvasive blood flow measurement.
  ABI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the ankle and arm.
  TBI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the toe and arm.
Period: Overall Study
Arm/Group | Healthy | Peripheral Artery Disease
Started | 52; 77 limbs | 143; 148 limbs
Completed | 52; 77 limbs | 83; 89 limbs
Not Completed | 0; 0 limbs | 60; 59 limbs

BASELINE CHARACTERISTICS:
Population: Site-reported demographic and medical history data are presented based on the assigned cohort using the definitions for Healthy and PAD (2) in the Groups and Interventions Section. Baseline information was not collected for one participant; therefore, a total of 194 participants were included in baseline analysis.
Units Other Than Participants: limbs
Groups:
- Peripheral Artery Disease (Including Critical Limb Ischemia): PAD cohort is all-comers to the vascular lab that are scheduled to undergo assessment for Peripheral Artery Disease (PAD) or have a planned endovascular or surgical intervention to address PAD.
  PAD (2) cohort patients are defined by ABI≤0.9 or ABI>1.4 and secondary verification of TBI≤0.7 without exhibition of symptoms and regardless of Rutherford Category. CLI cohort patients are defined by an exhibition of chronic rest pain and active wounds, verified by TBI<0.3. PAD (2) and CLI patients will receive FlowMet-R measurement in addition to their routine standard of care.
  FlowMet-R: FlowMet-R is a noninvasive blood flow measurement.
  ABI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the ankle and arm.
  TBI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the toe and arm.
- Total: Total of all reporting groups
Arm/Group | Healthy | Peripheral Artery Disease (Including Critical Limb Ischemia) | Total
Number analyzed (Participants) | 63 | 131 | 194
Number analyzed (limbs) | 77 | 148 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (13.0) | 70.4 (9.6) | 67.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 56 | 91
  Male | 28 | 75 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 32 | 36
  Not Hispanic or Latino | 59 | 99 | 158
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 21 | 26
  White | 55 | 78 | 133
  More than one race | NA — Not collected | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 2 | 31 | 33
Region of Enrollment [Number; unit: participants]
  United States | 63 | 131 | 194
Weight [Mean (Standard Deviation); unit: pounds] — Population: Data not collected for 4 healthy participants
  pounds
    number analyzed (Participants) | 59 | 131 | 190
    (all) | 183.4 (44.8) | 178.4 (42.6) | 180.5 (43.1)
Height [Mean (Standard Deviation); unit: inches] — Population: Data not collected for 4 healthy participants
  inches
    number analyzed (Participants) | 59 | 131 | 190
    (all) | 66.1 (4.1) | 66.5 (4.3) | 66.4 (4.2)
Body Mass Index [Mean (Standard Deviation); unit: lbs/(in^2)*703] — Population: Data not collected for 4 healthy participants
  lbs/(in^2)*703
    number analyzed (Participants) | 59 | 131 | 190
    (all) | 28.7 (7.3) | 28.2 (5.7) | 28.4 (6.3)
Medical History [Number; unit: participants]
  Chronic Obstructive Pulmonary Disease (COPD) | 3 | 24 | 27
  Type 1 diabetes | 2 | 3 | 5
  Type 2 diabetes | 18 | 65 | 83
  Clots or deep vein thrombosis (DVT) | 0 | 7 | 7
  Venous Disease | 12 | 35 | 47
Wound History [Count of Participants; unit: Participants] | 4 | 14 | 18
Smoking Status [Count of Participants; unit: Participants]
  Current | 5 | 31 | 36
  Previous | 24 | 67 | 91
  Never | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of FlowMet-R for Diagnosis of PAD and CLI
Description: Primary objective is to determine the efficacy of FlowMet-R measurements in diagnosing PAD & CLI. All patients were combined from healthy & PAD groups to form one cohort, ABI and TBI were then used to assign patients in PAD (1), PAD (2) & CLI. FlowMet-R data (comprised of blood flow measurements and/or feature analysis of the blood flow waveform) were used to create a predictive model of PAD severity. This model was used to generate diagnostic receiver operating characteristic (ROC) curves for PAD and, independently, CLI, at three time points.
  ROC curves were used to compute the peak sensitivity, peak specificity, and area under the curve (AUC) at the initial, 3-month and 6-month time points. Sensitivity, specificity and AUC are unitless. Sensitivity is the percentage of true positives & specificity is the percentage of true negatives at the location on the ROC curve where it was closest to the upper left of the unit square from an ROC curve (peak).
Time Frame: Initial, three month, and six month time points.
Population: Sensitivity, specificity and area under the curve (AUC) were calculated for PAD (1) vs. not PAD (1), PAD (2) vs not PAD (2), and CLI vs. not CLI at initial, three-month and six-month timepoints.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: limbs
Groups:
- Peripheral Artery Disease (1) vs Not PAD: All patients were assigned PAD (1) by the following criteria: ABI≤0.9 or ABI>1.4 and secondary verification of TBI≤0.7 with exhibition of at least mild claudication (Rutherford Category>0) and will receive FlowMet-R measurement in addition to their routine standard of care.
  FlowMet-R: FlowMet-R is a noninvasive blood flow measurement.
  ABI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the ankle and arm.
  TBI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the toe and arm.
  Not PAD are patients that did not meet the definition above.
- Peripheral Artery Disease (2) vs Not PAD: All patients were assigned PAD (2) by the following criteria: ABI≤0.9 or ABI>1.4 and secondary verification of TBI≤0.7 without exhibition of symptoms and will receive FlowMet-R measurement in addition to their routine standard of care.
  FlowMet-R: FlowMet-R is a noninvasive blood flow measurement.
  ABI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the ankle and arm.
  TBI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the toe and arm.
  Not PAD are patients that did not meet the definition above.
- Critical Limb Ischemia (CLI) vs Not CLI: All patients were assigned CLI based on exhibition of chronic rest pain and active wounds, verified by TBI<0.3. CLI cohort patients will receive FlowMet-R measurement in addition to their routine standard of care.
  FlowMet-R: FlowMet-R is a noninvasive blood flow measurement.
  ABI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the ankle and arm.
  TBI: Ankle Brachial Index is a ratio-metric blood pressure measurement in the toe and arm.
  Not CLI are patients that did not meet the definition above.
Arm/Group | Peripheral Artery Disease (1) vs Not PAD | Peripheral Artery Disease (2) vs Not PAD | Critical Limb Ischemia (CLI) vs Not CLI
Number analyzed (Participants) | 190 | 190 | 192
Number analyzed (limbs) | 218 | 218 | 220
probability
  Sensitivity (Initial) | 0.80 [0.73 to 0.87] | 0.78 [0.71 to 0.85] | 0.82 [0.66 to 0.98]
  Specificity (Initial) | 0.78 [0.70 to 0.87] | 0.86 [0.78 to 0.94] | 0.78 [0.72 to 0.84]
  Area Under the Curve (Initial) | 0.84 [0.78 to 0.89] | 0.87 [0.82 to 0.92] | 0.86 [0.80 to 0.93]
  Sensitivity (3 months): number analyzed (Participants) | 66 | 66 | 67
  Sensitivity (3 months): number analyzed (limbs) | 76 | 76 | 77
  Sensitivity (3 months) | 0.52 [0.38 to 0.67] | 0.57 [0.44 to 0.71] | 1.00 [1.00 to 1.00]
  Specificity (3 months): number analyzed (Participants) | 66 | 66 | 67
  Specificity (3 months): number analyzed (limbs) | 76 | 76 | 77
  Specificity (3 months) | 0.63 [0.46 to 0.81] | 0.77 [0.60 to 0.95] | 0.91 [0.84 to 0.97]
  Area Under the Curve (3 months): number analyzed (Participants) | 66 | 66 | 67
  Area Under the Curve (3 months): number analyzed (limbs) | 76 | 76 | 77
  Area Under the Curve (3 months) | 0.58 [0.45 to 0.71] | 0.67 [0.54 to 0.80] | 0.95 [0.86 to 1.00]
  Sensitivity (6 months): number analyzed (Participants) | 75 | 75 | 77
  Sensitivity (6 months): number analyzed (limbs) | 87 | 87 | 89
  Sensitivity (6 months) | 0.74 [0.62 to 0.86] | 0.73 [0.62 to 0.84] | 1.00 [1.00 to 1.00]
  Specificity (6 months): number analyzed (Participants) | 75 | 75 | 77
  Specificity (6 months): number analyzed (limbs) | 87 | 87 | 89
  Specificity (6 months) | 0.58 [0.41 to 0.74] | 0.67 [0.48 to 0.86] | 0.59 [0.48 to 0.69]
  Area Under the Curve (6 months): number analyzed (Participants) | 75 | 75 | 77
  Area Under the Curve (6 months): number analyzed (limbs) | 87 | 87 | 89
  Area Under the Curve (6 months) | 0.62 [0.49 to 0.74] | 0.67 [0.54 to 0.79] | 0.79 [0.39 to 1.00]

2. Secondary Outcome: Sensitivity and Specificity of FlowMet-R for Prognosis of Requiring a Peripheral Vascular Intervention
Description: ROC curves for predicting if a patient will undergo intervention following their initial visit were generated using FlowMet-R measurement data. ROC curves were used to compute the peak sensitivity, peak specificity, and area under the curve (AUC) within the 3-month and 6-month time points, separately. Sensitivity, specificity and AUC are unitless. Sensitivity is the percentage of true positives & specificity is the percentage of true negatives at the location on the ROC curve where it was closest to the upper left of the unit square from an ROC curve (peak).
Time Frame: Within three and six months following initial visit
Population: PAD (1), PAD (2) and CLI participants who underwent vascular intervention following their initial visit.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: limbs
Groups:
- Vascular Intervention Within 3 Months: Sensitivity, specificity and area under the curve (AUC) were calculated for PAD and CLI participants who underwent vascular reintervention within three-months following the initial visit.
- Vascular Intervention Within 6 Months: Sensitivity, specificity and area under the curve (AUC) were calculated for PAD and CLI participants who underwent vascular reintervention within six-months following the initial visit.
Arm/Group | Vascular Intervention Within 3 Months | Vascular Intervention Within 6 Months
Number analyzed (Participants) | 69 | 81
Number analyzed (limbs) | 80 | 92
probability
  Sensitivity | 0.60 [0.30 to 0.90] | 0.59 [0.35 to 0.82]
  Specificity | 0.49 [0.37 to 0.60] | 0.56 [0.45 to 0.67]
  Area Under the Curve (AUC) | 0.52 [0.32 to 0.71] | 0.54 [0.39 to 0.69]

3. Secondary Outcome: Sensitivity, Specificity and Area Under the Curve (AUC) of FlowMet-R in Diagnosing Significant Stenosis
Description: ROC curves for predicting a patient has significant stenosis, defined by greater than 50%, in at least one peripheral artery will be generated using FlowMet-R measurement data. ROC curves will be used to compute the peak sensitivity, peak specificity, and area under the curve (AUC) at the initial visit. Sensitivity, specificity and AUC are unitless. Sensitivity is the percentage of true positives & specificity is the percentage of true negatives at the location on the ROC curve where it was closest to the upper left of the unit square from an ROC curve (peak).
Time Frame: Initial visit
Population: All PAD participants with significant stenosis, defined by greater than 50%, in at least one peripheral artery and generated using FlowMet-R measurement data.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: limbs
Groups:
- PAD Participants With Significant Stenosis: All PAD participants with significant stenosis, defined by greater than 50%, in at least one peripheral artery and generated using FlowMet-R measurement data.
Arm/Group | PAD Participants With Significant Stenosis
Number analyzed (Participants) | 122
Number analyzed (limbs) | 134
probability
  Sensitivity | 0.61 [0.51 to 0.72]
  Specificity | 0.61 [0.48 to 0.75]
  Area Under the Curve (AUC) | 0.63 [0.53 to 0.73]

4. Secondary Outcome: Stenosis Percentage
Description: A correlation test will be performed between FlowMet-R and stenosis percentage.
  The correlations between the acceleration time from the FlowMet-R device and peripheral artery stenosis will be computed using a Pearson correlation. Correlation will be computed using available FlowMet-R data from PAD participants with significant stenosis, defined by greater than 50%, in at least one peripheral artery at the initial visit.
Time Frame: Initial visit
Population: All limbs of PAD participants with significant stenosis, defined by greater than 50%, in at least one peripheral artery and generated using FlowMet-R measurement data.
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Units Other Than Participants: limbs
Arm/Group | PAD Participants With Significant Stenosis
Number analyzed (Participants) | 122
Number analyzed (limbs) | 134
percentage of stenosis | 67.9 (32.5)
Statistical Analysis 1: Comparison: PAD Participants With Significant Stenosis; Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = 0.26, 95% CI 2-sided [0.10 to 0.41]

5. Secondary Outcome: Changes in Ankle Brachial Index (ABI)
Description: The outcome ABI is a ratio of blood pressures in the arm and ankle. Values less than 1 generally indicate narrower arteries. The outcome used the change in ABI for: 0 to 3 months, 0 to 6 months, and 3 to 6 months. The correlation with this outcome was estimated using the corresponding change in acceleration time from the FlowMet-R device.
Time Frame: Within three and six months following initial visit.
Population: Limbs of participants with ABI measured at 0, 3, and 6 months. ABI was not collected in at least 2 of the 86 limbs included in the overall analysis.
Measure: Mean (Standard Deviation); unit: mmHg / mmHg
Units Other Than Participants: limbs
Groups:
- 0 to 3 Months: Change in ABI between the initial and three-month follow-up visit.
- 0 to 6 Months: Change in ABI between the initial and six-month follow-up visit.
- 3 to 6 Months: Change in ABI between the three-month and six-month follow-up visits.
Arm/Group | 0 to 3 Months | 0 to 6 Months | 3 to 6 Months
Number analyzed (Participants) | 65 | 72 | 47
Number analyzed (limbs) | 75 | 84 | 57
mmHg / mmHg | 0.09 (0.23) | 0.08 (0.31) | 0.03 (0.22)
Statistical Analysis 1: Comparison: 0 to 3 Months; Correlation of change in acceleration time and ABI. Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = -0.26, 95% CI 2-sided [-0.46 to -0.03]
Statistical Analysis 2: Comparison: 0 to 6 Months; Correlation of change in acceleration time and ABI. Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = -0.33, 95% CI 2-sided [-0.51 to -0.12]
Statistical Analysis 3: Comparison: 3 to 6 Months; Correlation of change in acceleration time and ABI. Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = -0.13, 95% CI 2-sided [-0.38 to 0.14]

6. Secondary Outcome: Changes in Toe Brachial Index (TBI)
Description: The outcome TBI is a ratio of blood pressures in the arm and toe. Values less than 1 generally indicate narrower arteries. The outcome used the change in TBI for: 0 to 3 months, 0 to 6 months, and 3 to 6 months. The correlation with this outcome was estimated using the corresponding change in acceleration time from the FlowMet-R device.
Time Frame: Within three and six months following initial visit.
Population: Limbs of participants with TBI measured at 0, 3, and 6 months.
Measure: Mean (Standard Deviation); unit: mmHg / mmHg
Units Other Than Participants: limbs
Groups:
- 0 to 3 Months: Change in TBI between the initial and three-month follow-up visit.
- 0 to 6 Months: Change in TBI between the initial and six-month follow-up visit.
- 3 to 6 Months: Change in TBI between the three-month and six-month follow-up visits.
Arm/Group | 0 to 3 Months | 0 to 6 Months | 3 to 6 Months
Number analyzed (Participants) | 66 | 74 | 48
Number analyzed (limbs) | 76 | 86 | 58
mmHg / mmHg | 0.08 (0.24) | 0.10 (0.25) | 0.02 (0.18)
Statistical Analysis 1: Comparison: 0 to 3 Months; Correlation of change in acceleration time and TBI. Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = -0.34, 95% CI 2-sided [-0.52 to -0.12]
Statistical Analysis 2: Comparison: 0 to 6 Months; Correlation of change in acceleration time and TBI. Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = -0.35, 95% CI 2-sided [-0.52 to -0.15]
Statistical Analysis 3: Comparison: 3 to 6 Months; Correlation of change in acceleration time and TBI. Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = -0.24, 95% CI 2-sided [-0.47 to 0.02]

7. Secondary Outcome: Changes in Rutherford Classification
Description: Rutherford Classification is an ordinal scale that ranges from 0 to 6 and is used to measure peripheral arterial disease severity and chronic limb threatening ischemia. Higher values indicate more severe disease. The changes for Rutherford Classification were computed for: 0 to 3 months, 0 to 6 months, and 3 to 6 months. The correlation with this outcome was estimated using the corresponding change in acceleration time from the FlowMet-R device.
Time Frame: Within three and six months following initial visit.
Population: Limbs of participants with Rutherford Class measured at 0, 3, and 6 months. Rutherford Class was not collected in at least 2 of the 86 limbs included in the overall analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Groups:
- 0 to 3 Months: Change in Rutherford Classification between the initial and three-month follow-up visit.
- 0 to 6 Months: Change in Rutherford Classification between the initial and six-month follow-up visit.
- 3 to 6 Months: Change in Rutherford Classification between the three-month and six-month follow-up visits.
Arm/Group | 0 to 3 Months | 0 to 6 Months | 3 to 6 Months
Number analyzed (Participants) | 66 | 72 | 48
Number analyzed (limbs) | 76 | 84 | 58
units on a scale | -0.39 (1.4) | -0.62 (1.5) | -0.26 (1.2)
Statistical Analysis 1: Comparison: 0 to 3 Months; Correlation of change in acceleration time and Rutherford Classification. Descriptive analysis of endpoint with no hypothesis; Test type: Other; Correlation = 0.15, 95% CI 2-sided [-0.08 to 0.36]
Statistical Analysis 2: Comparison: 0 to 6 Months; [analysis description as in outcome 7, analysis 1]; Test type: Other; Correlation = 0.19, 95% CI 2-sided [-0.02 to 0.39]
Statistical Analysis 3: Comparison: 3 to 6 Months; [analysis description as in outcome 7, analysis 1]; Test type: Other; Correlation = 0.24, 95% CI 2-sided [-0.02 to 0.47]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the baseline assessment visit throughout 6-month follow-up.
Description: Investigators submitted device-related or suspected device-related AE or SAE to the sponsor and IRB within 5 business days after awareness. Sites were required to only include AEs that were reasonably associated with use of the FlowMet-R device. Investigators classified whether an AE was considered serious, non-serious and device related. All SAEs and AEs collected as part of the study are reported, including device- & non-device related events. All deaths reported on the Exit form are included.
Arm/Group | Healthy | Peripheral Artery Disease
All-Cause Mortality (participants affected / at risk) | 0/52 | 4/143
Serious Adverse Events (participants affected / at risk) | 0/52 | 6/143
Other Adverse Events (participants affected / at risk) | 0/52 | 2/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy (N=52) | Peripheral Artery Disease (N=143)
Amputation (Surgical and medical procedures) | 0 (0) | 3 (3)
Femoral Artery Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Femorofemoral Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Non-Healing Left Leg Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy (N=52) | Peripheral Artery Disease (N=143)
Pain during FlowMet-R Assessment (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Pain on first Digit due to device, temporarily removed device during procedure
Hematoma (Vascular disorders) | 0 (0) | 1 (1) — Hematoma in Left Groin

LIMITATIONS AND CAVEATS:
The study was terminated by Medtronic prior to completing enrollment. Difficulties with enrollment and limited compliance partially related to the COVID-19 pandemic limited the conclusions. Analyses described in the protocol were computed, but no hypothesis tests were completed. The AUC and its 95% CI are provided to assess the potential for the FlowMet device to classify CLI, PAD (1), PAD (2) at 0-, 3-, and 6-months, reintervention within 3- and 6-months, and significant stenosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT04120610/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT04120610/SAP_001.pdf